CLINICAL TRIAL: NCT02352922
Title: A Randomized Controlled Trial of Wound Infiltration With Extended-release Versus Short-acting Bupivacaine Before Laparoscopic or Robotic Hysterectomy
Brief Title: Randomized Trial of Wound Infiltration With Extended-release Bupivacaine Before Laparoscopic or Robotic Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 691275
Record Dates: First submitted 2015-01-27; First posted 2015-02-02 (Estimated); Results first posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Pain, Postoperative; Surgical Procedure, Unspecified
Keywords: Laparoscopy; Robotic Surgical Procedures; Hysterectomy; Anesthetics, Local; Bupivacaine; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liposomal Bupivacaine (Experimental): extended-release bupivacaine (EXPAREL)
  Interventions: Drug: Liposomal Bupivacaine
- Bupivacaine HCl (Active Comparator): short-acting bupivacaine
  Interventions: Drug: Bupivacaine HCl

INTERVENTIONS:
Drug: Liposomal Bupivacaine — pre-incision infiltration with liposomal bupivacaine
  Other Names: Exparel
  Arms: Liposomal Bupivacaine
Drug: Bupivacaine HCl — pre-incision infiltration with bupivacaine HCl
  Other Names: Marcaine
  Arms: Bupivacaine HCl

SUMMARY:
The investigators are studying ways to improve pain control after surgery. One way to decrease pain is to inject incisions with a numbing medicine (local anesthetic) while in the operating room. There is an FDA approved extended-release version of a commonly used local anesthetic (bupivacaine) that can last for 4 days instead of 6 hours. The investigators are studying whether using the extended-release medication (Exparel) will give better pain relief after laparoscopic and robotic-assisted hysterectomies.

DETAILED DESCRIPTION:
Lidocaine and bupivacaine hydrochloride (HCl) are the most commonly used drugs for wound infiltration during laparoscopic surgery for post-operative pain control. There is some evidence that wound infiltration decreases immediate post-operative pain. While bupivacaine has a slightly slower onset of action (5-10 minutes), it has become the preferred injectable anesthetic for surgical use because of its longer duration of effect (4-8 hours versus 1-2 hours for lidocaine).

DepoFoam bupivacaine (EXPAREL, Pacira Pharmaceuticals, Inc., Parsippany, NJ, USA) is a newer extended-release formulation of bupivacaine HCl approved by the U.S. Federal Drug Administration in October 2011. In this suspension, bupivacaine is encapsulated in microscopic spherical lipid-based particles of varying size to allow dispersion of the drug over an extended period of time. Analgesia is prolonged up to 96 hours. Given the extended duration of action, this liposomal bupivacaine may be better at providing post-operative pain relief in laparoscopic surgery.

Phase three trials have shown better pain control in the first 24 hours and less opioid use overall in bunionectomies, hemorrhoidectomies, and total knee replacement surgery when compared to placebo. No studies, however, have been published evaluating extended-release liposomal bupivacaine for laparoscopic surgery, or gynecologic surgery in general. Currently, we are using liposomal bupivacaine for pain relief after laparoscopic hysterectomies, but as stated, it has never been formally evaluated.

We hypothesize that liposomal bupivacaine ("extended-release") provides extended pain relief and decreases the need for supplemental opioid use after major laparoscopic surgery. We will be evaluating whether pre-incision infiltration of extended-release bupivacaine decreases post-operative pain from laparoscopic and robotic-assisted hysterectomy compared to bupivacaine HCl ("short-acting"). To achieve this evaluation we designed a double-blinded randomized controlled trial.

Patients who are scheduled to undergo a laparoscopic or robotic-assisted hysterectomy will be invited to participate. Group A will receive pre-incision infiltration of each trocar site with 4 ml of 0.25% Bupivacaine HCl. Group B will receive pre-incision infiltration of each trocar site with 4 ml of extended-release bupivacaine (EXPAREL) (13.3mg/ml). Subjects and outcome assessors will be blinded to group allocation.

Data will be collected while patients are in the hospital on pain levels and consumption of opioid pain medications. Upon discharge, pain levels, functioning, and quantity of opioid and non-steroidal anti-inflammatory (NSAID) pain medications will be collected through online questionnaires. Subjects will be followed until their 2-3 weeks post-operative visit.

ELIGIBILITY:
Inclusion Criteria:

1. Benign indication for surgery
2. Planned multiport laparoscopic or robotic assisted hysterectomy
3. Non-pregnant
4. Able to provide informed consent
5. Owns smartphone or computer with internet access
6. Willing to provide contact phone number and accept SMS text messages
7. Ability to speak and read English (because texts and online surveys will be in English only)

Exclusion Criteria:

1. Planned additional procedures (e.g. incontinence surgery, prolapse repair or bowel surgery)
2. Contraindication to study drug

   1. Severe Hepatic disease
   2. Severe Kidney disease
   3. Current use of monoamine oxidase inhibitors
   4. Current use of tricyclic antidepressants
3. History of substance or alcohol abuse within the past 2 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georgine Lamvu, MD, MPH, Principal Investigator — Florida Hospital Orlando; Kenneth I Barron, MD, Study Director — Florida Hospital Orlando
Locations (1):
- Florida Hospital Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
There is not a plan to make IPD available, but aggregate data can be made available to interested correspondents

REFERENCES:
- [Background] Saleh A, Fox G, Felemban A, Guerra C, Tulandi T. Effects of local bupivacaine instillation on pain after laparoscopy. J Am Assoc Gynecol Laparosc. 2001 May;8(2):203-6. doi: 10.1016/s1074-3804(05)60578-6. PMID 11342725
- [Background] Ke RW, Portera SG, Bagous W, Lincoln SR. A randomized, double-blinded trial of preemptive analgesia in laparoscopy. Obstet Gynecol. 1998 Dec;92(6):972-5. doi: 10.1016/s0029-7844(98)00303-2. PMID 9840560
- [Background] Loizides S, Gurusamy KS, Nagendran M, Rossi M, Guerrini GP, Davidson BR. Wound infiltration with local anaesthetic agents for laparoscopic cholecystectomy. Cochrane Database Syst Rev. 2014 Mar 12;2014(3):CD007049. doi: 10.1002/14651858.CD007049.pub2. PMID 24619479
- [Background] Bergese SD, Onel E, Portillo J. Evaluation of DepoFoam((R)) bupivacaine for the treatment of postsurgical pain. Pain Manag. 2011 Nov;1(6):539-47. doi: 10.2217/pmt.11.62. PMID 24645765
- [Background] Golf M, Daniels SE, Onel E. A phase 3, randomized, placebo-controlled trial of DepoFoam(R) bupivacaine (extended-release bupivacaine local analgesic) in bunionectomy. Adv Ther. 2011 Sep;28(9):776-88. doi: 10.1007/s12325-011-0052-y. Epub 2011 Aug 12. PMID 21842428
- [Background] Gorfine SR, Onel E, Patou G, Krivokapic ZV. Bupivacaine extended-release liposome injection for prolonged postsurgical analgesia in patients undergoing hemorrhoidectomy: a multicenter, randomized, double-blind, placebo-controlled trial. Dis Colon Rectum. 2011 Dec;54(12):1552-9. doi: 10.1097/DCR.0b013e318232d4c1. PMID 22067185
- [Background] Bramlett K, Onel E, Viscusi ER, Jones K. A randomized, double-blind, dose-ranging study comparing wound infiltration of DepoFoam bupivacaine, an extended-release liposomal bupivacaine, to bupivacaine HCl for postsurgical analgesia in total knee arthroplasty. Knee. 2012 Oct;19(5):530-6. doi: 10.1016/j.knee.2011.12.004. Epub 2012 Jan 28. PMID 22285545
- [Background] Kato J, Ogawa S, Katz J, Nagai H, Kashiwazaki M, Saeki H, Suzuki H. Effects of presurgical local infiltration of bupivacaine in the surgical field on postsurgical wound pain in laparoscopic gynecologic examinations: a possible preemptive analgesic effect. Clin J Pain. 2000 Mar;16(1):12-7. doi: 10.1097/00002508-200003000-00003. PMID 10741813

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Started | 32 | 32
Completed | 28 (completed POD14 Survey) | 28 (Completed POD14 survey)
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (8.6) | 45.4 (9.1) | 45.19 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 8 | 12
  White | 24 | 18 | 42
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 32 | 64
BMI [Mean (Full Range); unit: kg/m^2] | 29 [19.8 to 83.9] | 27.6 [19.3 to 43.7] | 28.3 [19.3 to 83.9]

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale (NRS) Post-operative Pain Score on Post-Operative Day 1 (POD1).
Description: Numerical Rating Scale (0-10) post-operative pain score on POD1, where 0 = no pain and 10 = worst pain imaginable
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 30 | 30
units on a scale | 4.17 (2.2) | 4.97 (2.6)

2. Secondary Outcome: NRS Pain Score at 2 Hours
Description: numeric rating scale (0-10), mean and SD, where 0 = no pain and 10 = worst pain imaginable
Time Frame: 2 hours post-op
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 30 | 31
units on a scale | 2.53 (2.53) | 2.74 (3.24)

3. Secondary Outcome: NRS Pain Score at 4 Hours
Description: Pain scale measured from 0-10, where 0 = no pain and 10 = worst pain imaginable
Time Frame: 4 hours post-op
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 30 | 31
Score on a scale | 3.87 (2.86) | 3 (2.95)

4. Secondary Outcome: NRS Pain Score at 8 Hours
Description: Pain scale (0-10), where 0 = no pain and 10 = worst pain imaginable
Time Frame: 8 hours post-op
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 30 | 30
Score on a scale | 3.77 (2.75) | 3.67 (3.01)

5. Secondary Outcome: NRS Pain Score at 16 Hours
Description: Pain scale (0-10), where 0 = no pain and 10 = worst pain imaginable
Time Frame: 16 hours post-op
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 29 | 29
score on a scale | 3.1 (3.18) | 3.97 (2.76)

6. Secondary Outcome: NRS Pain Score Post-op Day 2
Description: Pain scale (0-10), where 0 = no pain and 10 = worst pain imaginable
Time Frame: 2 days post-op
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 29 | 31
score on a scale | 3.34 (2.06) | 4.17 (2.16)

7. Secondary Outcome: NRS Pain Score Post-op Day 3
Description: Pain scale, where 0 = no pain and 10 = worst pain imaginable
Time Frame: 3 days post-op
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 29 | 30
score on a scale | 2.79 (2.26) | 4.07 (1.98)

8. Secondary Outcome: NRS Pain Score Post-op Day 14
Description: Pain scale (0-10), where 0 = no pain and 10 = worst pain imaginable
Time Frame: Post-Operative Day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 28 | 28
score on a scale | 1.64 (2.58) | 2.07 (2.58)

9. Secondary Outcome: Quality of Life as Measured by the Brief Pain Inventory (BPI)
Description: The brief pain inventory scale uses the 0 to 10 numerical rating scale to measure pain intensity under four different conditions. On the four conditions 0 = no pain, no relief, and does not interfere, whereas 10 = pain as bad as you can imagine, complete relief, and completely interferes
Time Frame: Post-Operative Day 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 29 | 31
score on a scale | 4.09 (2.58) | 4.31 (1.99)

10. Secondary Outcome: Quality of Life as Measured by the Brief Pain Inventory (BPI)
Description: as for outcome 9
Time Frame: Post-Operative Day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 29 | 30
score on a scale | 3.36 (2.71) | 3.94 (2.37)

11. Secondary Outcome: Quality of Life as Measured by the Brief Pain Inventory (BPI)
Description: at time of post-op visit The brief pain inventory scale uses the 0 to 10 numerical rating scale to measure pain intensity under four different conditions. On the four conditions 0 = no pain, no relief, and does not interfere, whereas 10 = pain as bad as you can imagine, complete relief, and completely interferes
Time Frame: Post-Operative Day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 28 | 28
score on a scale | 1.74 (2.61) | 1.65 (1.93)

12. Secondary Outcome: Total Opioid Use Prior to Hospital Discharge
Description: Oral morphine equivalent of opioid use while in the hospital
Time Frame: 24 hours
Measure: Mean (Full Range); unit: mg (oral morphine equivalents)
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 32 | 32
mg (oral morphine equivalents) | 216 [75 to 810] | 266 [54 to 634]

13. Secondary Outcome: Total Opioid Use End of Post-op Day 3
Description: Total use of home opioids by pill count/ oral morphine equivalents
Time Frame: 72 hrs post-op
Measure: Mean (Full Range); unit: mg (oral morphine equivalents)
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 29 | 30
mg (oral morphine equivalents) | 320 [115 to 766] | 344 [84 to 784]

14. Secondary Outcome: Total Opioid Use at Post-op Day 14
Description: Total use of home opioids by pill count/ oral morphine equivalents
Time Frame: Post-Operative Day 14
Measure: Mean (Full Range); unit: mg (oral morphine equivalents)
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 27 | 28
mg (oral morphine equivalents) | 360 [115 to 1086] | 443 [84 to 1234]

15. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: Post-Operative Day 14
Population: if a patient reported a particular adverse effect at more than one time point, the patient was counted only once. Patients may report more than one adverse effect. Analysis and percentages reflect only those with complaints of adverse effects.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
Number analyzed (Participants) | 16 | 25
Participants
  Gas distension/bloated | 5 | 9
  Constipation | 5 | 2
  Nausea | 4 | 6
  Headache | 2 | 7
  Sore throat/cough | 1 | 3
  Dizziness | 1 | 3

ADVERSE EVENTS:
Arm/Group | Liposomal Bupivacaine | Bupivacaine HCl
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

LIMITATIONS AND CAVEATS:
study published in JMIG. https://doi.org/10.1016/j.jmig.2016.11.002

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No